CLINICAL TRIAL: NCT06241339
Title: Chronic Effect of Mat Pilates on Neuromotor, Cardiovascular Functions and Inflammatory Markers in Individuals Post-Stroke Stroke and High Blood Pressure
Status: Available | Type: Expanded Access
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Postgraduate scholarship (Unknown)
Responsible Party: Principal Investigator, Jeferson Silva da Rocha, teacher, Rio de Janeiro State University
Other Study IDs: 69237423.2.0000.5259
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Stroke; High Blood Pressure
Keywords: Autonomy; hemodynamic; balance; muscle strength; chronic reduction in blood pressure
MeSH Terms: conditions — Stroke; Hypertension

INTERVENTIONS:
Other: Mat Pilates — Mat Pilates training will last 12 weeks, with three weekly trial sessions being held at 48-72h intervals. Each session will last approximately 60 minutes, including: 5 minutes of warm-up (light calisthenic exercises for the shoulder and pelvic girdles); 50 minutes of Mat Pilates exercises; 5 min back to calm.
  Upon arriving at the training site, volunteers will rest for 10 minutes in a sitting position, after which BP measurements will be taken and HR at rest. Throughout consecutive training sessions, participants will perform Pilates method exercises with a progressively greater degree of difficulty and complexity, following the official recommendations for prescription of resistance exercise for individuals with BP elevated and post-stroke. The exercises will be performed in single sets of 10 repetitions. Groups will be advised to maintain daily activities without physical exercise during the 12-week period.

SUMMARY:
The Pilates method aims to develop conscious control of body movements. In the literature there are studies that relate the method to postural stabilization, joint rehabilitation, treatment of low back pain, cancer and chronic obstructive pulmonary disease. However, studies on the modality's potential for improving isokinetic and antihypertensive strength are scarce, particularly in post-stroke hemiparetic individuals with high blood pressure (BP). The objective of the study is to investigate changes in isokinetic strength and BP, in addition to functional capacity, balance, autonomic modulation, blood biomarkers and endothelial function in hemiparetic individuals due to stroke sequelae and/or with high BP (prehypertensive and hypertensive), after 12 weeks of training with Mat Pilates. Eligible volunteers will be randomly divided into a Mat Pilates group with stroke (GP-AVE), Mat Pilates group with high blood pressure (HA) (GP-HA), control group with stroke (GC-AVE) and control group with HA (GC-HA ). On the first and second visit, measurements of isokinetic strength, functional capacity, static and dynamic balance, heart rate variability, cardiac output, stroke volume, endothelial function, total peripheral vascular resistance and blood biomarkers will be carried out. In addition, 24-hour BP will be measured by ambulatory monitoring (ABPM). GP-AVE and GP-HA will participate in a 12-week Mat Pilates program, totaling 36 training sessions lasting approximately 60 minutes, with an increasing degree of difficulty and complexity throughout the training period. GC-AVE and GC-HA will be instructed to maintain their daily activities during the intervention period, then they will be invited to participate in the Mat Pilates program. The initial measurements will be repeated at the end of the intervention in the Mat Pilates and control groups. Intra and intergroup comparisons will be carried out for all outcomes, for a significance level set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria: Hemiparetic individuals with a history of stroke and/or high blood pressure (prehypertensive and hypertensive patients) who are controlled and do not practice the Pilates method.

Exclusion Criteria: Diagnosis of cardiovascular, respiratory, metabolic or locomotor disease that makes it impossible or contraindicates the practice of the proposed exercises; Uncontrolled hypertension (systolic BP ≥160 mmHg or diastolic pressure and ≥105 mmHg at rest); Spasticity: 3 according to the modified Ashworth Scale; Smoking and frequencies in exercise sessions below 75%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Jeferson Silva da Rocha, Rio de Janeiro, Brazil